CLINICAL TRIAL: NCT07393646
Title: Prospective Evaluation of a Digital Health and Telephonic Coaching Program for Health Prevention
Brief Title: Digital Prevention Program With Telephonic Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivoptim Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VIVOPTIM-DH-2015
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Risk; Cardiovascular Disease Prevention; Health Behavior Change; Lifestyle (Sedentary Behavior and Physical Activity); Lifestyle Risk Reduction
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital and Telephonic Prevention Program (Experimental): Participants received access to a digital prevention platform with personalized content and educational resources. They also received regular structured telephonic support from trained healthcare professionals, including coaching and behavioral guidance to improve lifestyle factors such as physical activity, diet, and cardiovascular risk management. All participants were assigned to this intervention without randomization or control group.
  Interventions: Behavioral: Digital Health Platform; Behavioral: Telephonic Coaching

INTERVENTIONS:
Behavioral: Digital Health Platform — Customized digital platform providing educational content, tools, and resources to support lifestyle changes and improve cardiovascular risk factors, including diet and physical activity. Participants had access to personalized dashboards and tracking features.
Behavioral: Telephonic Coaching — Structured telephonic support provided by trained healthcare professionals. Includes regular calls to provide guidance, monitor progress, support behavior change, and reinforce adherence to healthy lifestyle interventions.

SUMMARY:
This study evaluates a digital health prevention program combining digital tools and structured telephonic coaching to support adult participants in improving health-related behaviors and well-being.

Participants voluntarily enrolled in an ongoing prevention program offering personalized digital content, educational resources, and regular telephone-based support provided by trained professionals. The program aims to promote healthier lifestyles, prevent the development of chronic conditions, and improve overall health outcomes.

The study analyzes data collected from a defined cohort of participants enrolled during a specific period to assess changes in health-related outcomes, engagement, and adherence to the program. The results are intended to contribute to the evidence base for digital and telephonic prevention interventions in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Voluntary enrollment in the digital prevention program.
* Access to digital devices (computer, tablet, or smartphone) to use the digital platform.
* Consent to participate in the program and allow the use of data for research purposes.
* For the analysis cohort: at least one year of participation in the program.
* Insured people of MGEN health insurance

Exclusion Criteria:

* Participants who did not provide consent for the use of their data in research.
* Participants with incomplete baseline cardiovascular risk data.
* Participants who withdrew from the program before one year of participation.
* Participants without follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2688 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Change in Global Cardiovascular Risk Level (GCRL) | 1 year, 2 years or more (from program enrollment)
  The primary outcome is the change in participants' Global Cardiovascular Risk Level (GCRL), assessed on a 3-level scale (1: low, 2: medium, 3: high) at inclusion and at yearly follow-up. Improvement is defined as a decrease by at least one level in GCRL, deterioration as an increase by at least one level in GCRL and stable for a constant GCRL

SECONDARY OUTCOMES:
Physical Activity Level | 1 year, 2 years or more
  The proportion of participants meeting recommended physical activity levels, assessed at baseline and yearly follow-up. Changes over time are analyzed to determine behavioral improvements associated with program use.
Dietary Habits - Mediterranean Diet Adherence | 1 year, 2 years or more
  The proportion of participants adhering to a Mediterranean diet, assessed at baseline and yearly follow-up. Changes over time are analyzed to determine behavioral improvements associated with program use.
Duration of program participation | 1 year, 2 years and more than 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Vivoptim Solutions, Paris, France

IPD SHARING:
Plan to Share IPD: No